CLINICAL TRIAL: NCT06937840
Title: Comparison of Optimal Endotracheal Tube Depth Using Four Different Formulas (Based on Age, Height, Weight, and Third Finger Length) in Children Aged 1-4 Years and Verification With Fiberoptic Bronchoscopy
Brief Title: Comparison of Optimal Endotracheal Tube Depth Using Four Different Formulas in Children Aged 1-4 Years and Verification With Fiberoptic Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ozlem Can, Professor, Ankara University
Other Study IDs: AU-AR-OC-03
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Surgical Procedures Requiring Endotracheal Intubation Under General Anesthesia
Keywords: Pediatric airway, endotracheal tube, intubation depth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
. The optimal position of the endotracheal tube (ETT) within the trachea is the middle third portion, distal to the vocal cords. In addition to clinical assessments, methods such as posteroanterior chest radiography (PA-CXR) and fiberoptic bronchoscopy (FOB) can be used to verify ETT placement.

In our study, we aim to explain the relationship between the most accurate endotracheal tube depth and various formulas by using fiberoptic bronchoscopy, with the help of four different formulas based on age, height, weight, and third finger length.The study further seeks to:

1. To identify the most accurate formula for estimating ETT placement depth in the pediatric population living in Turkey.
2. To reduce the potential complications that may arise from incorrect ETT depth.
3. To determine which formula, when verified by fiberoptic bronchoscopy, is also consistent with auscultation findings-especially in situations where chest radiography or fiberoptic bronchoscopy may not be readily available.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 , 2 or 3
* Patients scheduled for elective surgical procedures
* Informed consent must be obtained from both the patient and, if applicable, their parent or guardian.

Exclusion Criteria:

* Patients under 1 year old or over 4 years old
* Patients with tracheobronchial anomalies
* Patients with vertebral column anomalies
* Patients with a history of tracheostomy and difficult intubation
* Patients who do not want to be included in the study
* Children with finger anomalies and syndromic associations
* Cases requiring nasal intubation

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Between 1 and 4years of ages pediatric patients scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the correct depth of endotracheal tube insertion | only once
  This study aims to identify the optimal endotracheal tube insertion depth in pediatric patients by evaluating tracheal dimensions using fiberoptic bronchoscopy.
A comparative analysis of four formulas used to determine endotracheal tube positioning | only once
  This study aims to identify the most accurate formula for estimating the ideal endotracheal tube depth among those based on age, weight, height, and middle finger length."

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided